CLINICAL TRIAL: NCT04328610
Title: A Randomized Controlled Trial to Assess the Efficacy of the Lymphatic Microsurgical Preventive Healing Approach (LYMPHA) to Prevent Lymphedema After Axillary Dissection for Breast Cancer
Brief Title: To Assess the Efficacy of the LYMPHA in the Prevention of Lymphedema Following Axillary Dissection for Breast Cancer
Acronym: LYMPHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1912-010-086
Record Dates: First submitted 2020-03-29; First posted 2020-03-31 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Lymphedema, Breast Cancer
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYMPHA technique group (Experimental): LVA at the time of Axillary Dissection
  Interventions: Procedure: LYMPHA(LYmphatic Microsurgical Preventive Healing Approach) technique
- Non-LYMPHA technique group (No Intervention): No preventive surgical approach

INTERVENTIONS:
Procedure: LYMPHA(LYmphatic Microsurgical Preventive Healing Approach) technique — Patients will receive a lymphatic-venous anastomosis at time of their required Axillary Dissection
  Arms: LYMPHA technique group

SUMMARY:
Lymphedema is the Build-up of Lymph Fluid in the Body's Tissue Causing Chronic, Debilitating Swelling. This Commonly Occurs as a Result of a Disruption of the Lymphatic System During Lymph Node Dissection Surgeries. LYMPHA (LYmphatic Microsurgical Preventive Healing Approach) is an Innovative Microsurgical Technique Where Blocked Lymphatic Vessels Are Drained Into the Blood Circulation by Surgically Creating a Shunt Between a Lymphatic Channel and a Blood Vessel Called a Lymphatic-venous Bypass. Recently, LYMPHA Technique Has Been Shown to Prevent Lymphedema When Performed at the Time of Nodal Dissection. We Propose a Prospective Study Evaluating the Effectiveness of LYMPHA Technique Using Objective Clinical Protocol.

DETAILED DESCRIPTION:
Consenting patients will have the LYMPHA procedure at the time of planned axillary dissection surgery for the prevention of upper and extremity lymphedema. The node dissection will be performed by Dr. Kang while the LYMPHA technique will be performed by the plastic surgeon, Dr. Kim. The LYMPHA procedure consist of performing LVA at the time of the node dissection. Patent blue dye will be injected in the volar surface of the upper third of the arm in a quantity of about 1-2 ml intradermally, subcutaneously, and under muscular fascia into patient approximately 10 minutes before skin incision. This will allow mapping of the lymphatic channels for identification for bypass. The node dissection will then be performed with preservation of the anterior branch of the axillary vein in the axilla. Afferent lymphatic vessels will be sutured into a branch of the axillary vein distal to a competen valve. The total duration of the surgery is approximately 3 hours. The LYMPHA technique accounts for an additional 30 min to the standard 2-2.5 hours allocated to the node dissection.

Pre-surgery, patients will have baseline limb circumference measurements of both the surgery-affected and unaffected arms and by lymphoscintigraphy. Patients will be followed up clinically at every 6 months up to a year. At each follow-up visit, patients will have a physical examination and their circumference of their limbs taken. Patients will also fill out a LyQLI, SF-36, DASH administered by the Clinical Research Coordinator pre-and post-surgery. Each patient will have a total of 1 years of participation time.

ELIGIBILITY:
Inclusion Criteria:

* Node-positive cancer requiring an axillary or lymphadenectomy
* Below 30 Body Mass Index

Exclusion Criteria:

* Patients receiving a sentinel lymph node biopsy
* Patients with established preoperative lymphedema
* Patients with post-thrombotic syndrome, peripheral vascular disease
* Pregnant patients

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
lymphatic flow | 6 months
  Difference in lymphatic flow between LYMPHA technique group and Non-LYMPHA technique group
limb volume | 6 months
  Difference in limb volume between LYMPHA technique group and Non-LYMPHA technique group
lymphatic flow | 1 year
  Difference in lymphatic flow between LYMPHA technique group and Non-LYMPHA technique group
limb volume | 1 year
  Difference in limb volume between LYMPHA technique group and Non-LYMPHA technique group

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, Seo-Gu, South Korea